CLINICAL TRIAL: NCT05505656
Title: Accuracy of Endomyometrial Biopsy in Diagnosis of Adenomyosis. A Prospective Cross-sectional Study
Brief Title: Accuracy of Endomyometrial Biopsy in Diagnosis of Adenomyosis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, Professor of Obstetrics and Gynecology, Ain Shams University
Other Study IDs: MD 129/ 2022
Record Dates: First submitted 2022-08-14; First posted 2022-08-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: hysteroscopic guided endomyometrial biopsy — we will obtain hysteroscopic guided endomyometrial biopsy in cases of adenomyosis

SUMMARY:
This study will compare the accuracy of diagnosing adenomyosis by obtaining hysteroscopic guided endomyometrial biopsy and comparing it to accuracy of diagnosis by transvaginal ultrasound and magnetic resonance imaging.

DETAILED DESCRIPTION:
Preoperative diagnosis of adenomyosis is usually difficult. The use of ultrasound and MRI for preoperative diagnosis is still of low positive predictive values. The majority of cases of adenomyosis are diagnosed postoperatively after justo pathological examination of the hysterectomy specimens.

The introduction of the concept of preoperative diagnosis of adenomyosis through a hysteroscopic endomyometrial biopsies may be a very good method for preoperative diagnosis of this condition. Participants patients who are diagnosed as adenomyosis by Ultrasound and MRI and scheduled for hysterectomy will undergo an endomyometrial biopsy. The accuracy of this method, its sensitivity, specificity, positive and negative predictive values of this method will be compared with the conventional methods for preoperative diagnosis of adenomyosis after final diagnosis by final gusto pathological diagnosis of hysterectomy specimens.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with abnormal uterine bleeding due to adenomyosis diagnosed by transvaginal ultrasound and mri and scheduled for hysterectomy

Exclusion Criteria:

* hysterectomy not performed
* incomplete ultrasound and mri information

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with abnormal uterine bleeding as diagnosed by ultrasound and mri
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
To compare endomyometrial biopsy with postoperative pathology to calculate Accuracy and likelihood ratio of endomyometrial biopsy to diagnose adenomyosis . | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive values of endomyometrial biopsy for diagnosis of adenomyosis compared to US and MRI | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Laban, Principal Investigator — Professor of Obstetrics and Gynecology
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided